CLINICAL TRIAL: NCT04392622
Title: A Phase I Study of d-Limonene With Concurrent Radiation and Platinum Based Chemotherapy for Xerostomia Prevention in Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: d-Limonene +Radiation +PlatinumBasedChemo for Xerostomia Prevention in LocallyAdvanced HNSCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-51656; 1P01CA257907-01A1 (NIH); NCI-2021-03256 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia | interventions — Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- d-limonene -2gram (Experimental): 2 gram d-limonene orally, once daily delivered during chemoradiation
  Interventions: Drug: D-Limonene Gelcaps; Radiation: Intensity modulated radiotherapy (IMRT); Drug: Cisplatin; Other: Xerostomia questionnaire
- d-limonene -4gram (Experimental): 4 gram d-limonene orally, as 2 grams 2 times daily delivered during chemoradiation
  Interventions: Drug: D-Limonene Gelcaps; Radiation: Intensity modulated radiotherapy (IMRT); Drug: Cisplatin; Other: Xerostomia questionnaire
- d-limonene -6gram (Experimental): 6 gram d-limonene orally, as 3 grams 2 times daily delivered during chemoradiation
  Interventions: Drug: D-Limonene Gelcaps; Radiation: Intensity modulated radiotherapy (IMRT); Drug: Cisplatin; Other: Xerostomia questionnaire
- d-limonene -8gram (Experimental): 8 gram d-limonene orally, as 4 grams 2 times daily delivered during chemoradiation
  Interventions: Drug: D-Limonene Gelcaps; Radiation: Intensity modulated radiotherapy (IMRT); Drug: Cisplatin; Other: Xerostomia questionnaire
- de-escalation dose d-limonene -6gram (Experimental): 6 gram d-limonene orally, as 3 grams 2 times daily delivered during chemoradiation
  Interventions: Drug: D-Limonene Gelcaps; Radiation: Intensity modulated radiotherapy (IMRT); Drug: Cisplatin; Other: Xerostomia questionnaire
- de-escalation dose d-limonene -4gram (Experimental): 4 gram d-limonene orally, as 2 grams 2 times daily delivered during chemoradiation
  Interventions: Drug: D-Limonene Gelcaps; Radiation: Intensity modulated radiotherapy (IMRT); Drug: Cisplatin; Other: Xerostomia questionnaire
- de-escalation dose d-limonene -2gram (Experimental): 2 gram d-limonene orally, once daily delivered during chemoradiation
  Interventions: Drug: D-Limonene Gelcaps; Radiation: Intensity modulated radiotherapy (IMRT); Drug: Cisplatin; Other: Xerostomia questionnaire

INTERVENTIONS:
Drug: D-Limonene Gelcaps — Administered orally at 2 to 8 grams daily
Radiation: Intensity modulated radiotherapy (IMRT) — Standard of Care -All patients will receive standard radiation treatment of 66 to 70 Gy given in 33 to 35 fractions (2 to 2.12 Gy/fractions) over 6.5 to 7 weeks.
Drug: Cisplatin — Standard of Care -Cisplatin as 100 mg/m2 IV
Other: Xerostomia questionnaire — Xerostomia questionnaire consists of 4 items on dryness while eating/speaking and 4 on dryness at rest. Patients rate each symptom on an 11 point ordinal Likert scale from 0 to 10, with higher scores indicating greater xerostomia

SUMMARY:
This study explores the safety of d-limonene, a commercially-available dietary supplement (food) as a potential therapeutic for the severe dry mouth (xerostomia) experienced by patients with head and neck cancer as a side effect of their anti-cancer treatment.

DETAILED DESCRIPTION:
Primary Objective:To determine the maximum tolerated dose (MTD) of d limonene when combined with radiation and platinum based chemotherapy in subjects with loco regionally advanced head and neck squamous cell carcinoma (HNSCC) based upon dose limiting toxicity (DLT)

Secondary Objective:

* To evaluate the feasibility and subject compliance with adjuvant administration of d limonene daily up to a maximum of 4 months after completion of chemoradiation
* To correlate the level of d-limonene measured in the plasma to the dose levels(s) administered to the subject
* To correlate the level of d limonene measured in the plasma to saliva flow rate and xerostomia questionnaire scores in subjects enrolled in this trial

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced loco regional squamous cell carcinoma of the nasopharynx (AJCC v8 Stage II IV); oropharynx (AJCC v8 Stage I III for HPV+ cancer, excluding T1 2N0; AJCC v8 Stage III IV for Human papillomavirus (HPV) negative cancer); larynx (AJCC v8 Stage III to IV); or hypopharynx (AJCC v8 Stage III to IV), scheduled to undergo chemoradiation. Patients with squamous cell carcinoma of the head and neck from an unknown primary site with involved nodes (N1 to 3) also qualify.
* Scheduled to received definitive RT with concurrent platinum based chemotherapy at Stanford
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 1
* Must be able to swallow d limonene gelcaps at the time of enrollment.
* Adequate hepatic function within 2 weeks prior to registration defined as follows: Bilirubin ≤ 2 mg/dL; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 times the upper limit of normal
* Adequate hematologic function within 2 weeks prior to registration defined as follows:

  * Absolute neutrophil count (ANC): ≥ 1,500/mm3
  * Platelets: ≥ 100,000/mm3
  * Hemoglobin: ≥ 8.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dL is acceptable).
* Adequate renal function defined as follows:

Serum creatinine ≤ 1.5 mg/dL within 2 weeks prior to registration or creatinine clearance (CC) ≥ 50 mL/min within 2 weeks prior to registration determined by 24 hour collection or estimated by Cockcroft Gault formula:

CCr male = [(140 - age) x (wt in kg)] [(Serum Cr mg/dL) x (72)] CCr female = 0.85 x (CrCl male)

* Negative serum pregnancy test within 2 weeks prior to registration and agreement to use a birth control method during the entire duration of d limonene treatment for women of childbearing potential
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of allergic reactions attributed to citrus fruits
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Dose limiting Toxicity | 9 weeks
  Dose limiting toxicity is defined as d-limonene related toxicity causing:
  * Greater than 1 week delay in completing the radiation course.
  * Inability to receive ≥ 66 Gy of radiotherapy.
  * Inability to receive at least 200 mg/m2 of total cisplatin equivalent dose or a total area under the curve (AUC) of 10 for carboplatin equivalent dose due to toxicity related to d-limonene Grade 3 or higher diarrhea that is attributable to the study drug.
  * Grade 3 abdominal pain that is attributable to the study drug. The outcome will be reported as the number of participants per dose level who experience any DLT (a number without dispersion / variance).

SECONDARY OUTCOMES:
Feasibility of adjuvant d-limonene administration | 4 months
  Participant compliance with adjuvant administration of d-limonene will be assessed as completing at least 14 weeks of per protocol adjuvant d-limonene treatment. The outcome is reported as the number of participants per dose level that were compliant.
Xerostomia toxicity | 12 months post completion of chemoradiation
  The degree of xerostomia will be assessed by the xerostomia survey. The survey consists of 8 items: 4 items regarding dryness or discomfort while eating or chewing and 4 items regarding dryness and discomfort while not eating or chewing. The participant will rate each item on a Likert scale from 0 to 10 (least effect to most severe effect) with higher scores implying greater dryness or discomfort. A summary score is calculated by summing the scores for each item and linearly transforming the score to produce a final score on a scale from 0 to 100. The outcome is reported as the mean and standard deviation of the final transformed scores from all subjects with survey results, by treatment level.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No